CLINICAL TRIAL: NCT05155449
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effect of Probiotics on Gut Function in Healthy Chinese Adults
Brief Title: Probiotic Intervention for Gut Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC19132
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gut Function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics (Active Comparator): Two capsules per day for 8 weeks
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Two capsules per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Capsule
  Arms: Probiotics
Dietary Supplement: Placebo — Capsule
  Arms: Placebo

SUMMARY:
The effect of probiotics on gut function in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* BMI between 18.5 and 27.9 kg/m²
* Subjects having ≥ 3 bowel movements per day
* Subject not satisfied with their bowel habits
* Subject having frequent stools during more than 4 weeks
* For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study
* Subjects agreeing to keep their dietary and life habits unchanged throughout the study
* Good general and mental health within the opinion of the investigator
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by a dated and signed ICF

Exclusion Criteria:

* Suffering IBS according to Rome IV criteria, chronic intestinal disease, immunodeficiency disorder or immunosuppressive treatment
* Clinically significant frequent constipation or diarrhea at the screening visit as judged by the Investigator
* Suffering from a severe chronic disease or GI disorders found to be inconsistent with the conduct of the study by the investigator
* Intake of antibiotics within 8 weeks prior to the start of the study
* With regular intake of probiotics within four weeks prior to V1 visit
* Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the V1 visit
* Suspected alcohol or substance abuse
* Use of medications other than contraceptives or prescribed medication after consulting with the investigator
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk if participating in the study, or influence the results or the subject´s ability to participate in the study
* With a known gluten intolerance, milk protein allergy
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredients
* Pregnant or lactating women or intending to become pregnant within 3 months ahead
* With significant change in food habits or in physical activity in the 3 months before the V1 visit
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator
* Having a lifestyle deemed incompatible with the study according to the investigator
* Currently participating in another clinical study, has done so in the past 30 days or being in the exclusion period of a previous clinical trial
* Under legal protection (guardianship, wardship) or deprived from his/her rights following administrative or judicial decision
* Presenting a psychological or linguistic incapability to sign the informed consent or Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements
* Impossible to contact in case of emergency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Bowel movements | 8 weeks
  Reduction of the number of bowel movements

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Meng, MD, Principal Investigator — Shanghai 9th People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Shanghai 9th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No